CLINICAL TRIAL: NCT01005550
Title: Determining the Minimum Effective Ropivacaine Dose for Unilateral Hypobaric Spinal Anaesthesia During Traumatic Femoral Neck Surgery in the Aged Person: Prospective Comparative Randomized Study
Brief Title: Ropivacaine Hypobaric Spinal Anaesthesia in Traumatic Hip Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2008.519
Record Dates: First submitted 2009-08-14; First posted 2009-11-02 (Estimated); Last update posted 2019-05-28 (Actual); Status verified 2010-12

CONDITIONS: Femoral Neck Fracture
Keywords: Unilateral spinal anaesthesia; Hypobaric anaesthesia; Ropivacaine; Traumatic hip surgery
MeSH Terms: conditions — Femoral Neck Fractures | interventions — Ropivacaine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- 6 mg of ropivacaine (Experimental): 6 mg of ropivacaine are used for the spinal anaesthesia
  Interventions: Drug: 6 mg of ropivacaine
- 8 mg of ropivacaine (Experimental): 8 mg of ropivacaine are used for the spinal anaesthesia
  Interventions: Drug: 8 mg of ropivacaine
- 10 mg of ropivacaine (Experimental): 10 mg of ropivacaine are used for the spinal anaesthesia
  Interventions: Drug: 10 mg of ropivacaine
- 12 mg of ropivacaine (Experimental): 12 mg of ropivacaine are used for the spinal anaesthesia
  Interventions: Drug: 12 mg of ropivacaine

INTERVENTIONS:
Drug: 6 mg of ropivacaine — 6 mg of ropivacaine are used for the spinal anaesthesia
  Arms: 6 mg of ropivacaine
Drug: 8 mg of ropivacaine — 8 mg of ropivacaine are used for the spinal anaesthesia
  Arms: 8 mg of ropivacaine
Drug: 10 mg of ropivacaine — 10 mg of ropivacaine for the spinal anaesthesia
  Arms: 10 mg of ropivacaine
Drug: 12 mg of ropivacaine — 12 mg of ropivacaine for the spinal anaesthesia
  Arms: 12 mg of ropivacaine

SUMMARY:
This is a prospective, monocentric, randomized study, comparing the effectiveness and tolerance of four different dosages of hypobaric ropivacaine for unilateral spinal anaesthesia during traumatic femoral neck surgery in the elderly.

ELIGIBILITY:
Inclusion Criteria:

* older than 70
* dorsal decubitus surgery
* ASA score 1, 2, 3
* MMS score > or equal to 25

Exclusion Criteria:

* local anesthetic allergy
* spinal anaesthetic exclusion
* MMS score lower than 25

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 64 (Actual)
Dates: Start 2009-04; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Determine the minimum effective ropivacaine dose for unilateral hypobaric spinal anaesthesia during traumatic femoral neck surgery. | 1 hour (surgery intervention)

SECONDARY OUTCOMES:
Spinal anaesthesia characteristics | 1 hour (surgery intervention)
Hemodynamics consequences | 1 hour (surgery intervention)
Patient and surgeon satisfaction | 1 hour (surgery intervention)
Morbidity and mortality | During 3 days after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Pascal MEURET, MD, Principal Investigator — Hospices Civils de Lyon
Locations (1):
- Hospices Civils de Lyon, Lyon, France

REFERENCES:
- [Result] Lilot M, Meuret P, Bouvet L, Caruso L, Dabouz R, Deleat-Besson R, Rousselet B, Thouverez B, Zadam A, Allaouchiche B, Boselli E. Hypobaric spinal anesthesia with ropivacaine plus sufentanil for traumatic femoral neck surgery in the elderly: a dose-response study. Anesth Analg. 2013 Jul;117(1):259-64. doi: 10.1213/ANE.0b013e31828f29f8. Epub 2013 Apr 16. PMID 23592605